CLINICAL TRIAL: NCT03515434
Title: The Effectiveness of Erector Spinae Plane Block and Transversus Abdominis Plane Block for Postoperative Analgesia in Inguinal Hernia Repair Undergoing Spinal Anesthesia
Brief Title: Comparison of Transversus Abdominis Plane Block and Erector Spinae Plane Block in Inguinal Hernia Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maltepe University (Other)
Responsible Party: Principal Investigator, Asst. Prof. Serkan Tulgar, M.D., assiatant proffessor, Maltepe University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: TAPvsESP
Record Dates: First submitted 2018-04-21; First posted 2018-05-03 (Actual); Last update posted 2018-05-24 (Actual); Status verified 2018-05

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ESP Block (Active Comparator): Ultrasound-guided Erector spinae plane (ESP) block will be performed at the finishing of the surgery with 30 ml of a bupivacaine/lidocaine mixture. The postoperative routine analgesic protocol will be performed (consist of intravenous analgesics and intravenous patient-controlled analgesia) with no additional intervention (block) Standard Pain Followup and Monitorization will be performed
  Interventions: Procedure: ESP Block; Other: Standard Pain Followup and Monitorization
- TAP Block (Active Comparator): Ultrasound-guided Transversus abdominis plane (TAP) block will be performed at the finishing of the surgery with 30 ml of a bupivacaine/lidocaine mixture. The postoperative routine analgesic protocol will be performed (consist of intravenous analgesics and intravenous patient-controlled analgesia) with no additional intervention (block) Standard Pain Followup and Monitorization will be performed
  Interventions: Procedure: TAP Block
- Control (Sham Comparator): The postoperative routine analgesic protocol will be performed (consist of intravenous analgesics and intravenous patient-controlled analgesia) with no additional intervention (block) Standard Pain Followup and Monitorization will be performed.
  Interventions: Other: Standard Pain Followup and Monitorization

INTERVENTIONS:
Procedure: ESP Block — ESP block will be performed at the finishing of surgery under spinal anesthesia. A convex ultrasound transducer will be placed in a longitudinal parasagittal orientation 2-3 cm lateral to T10 spinous process. The erector spinae muscles will be identified superficial to the tip of T10 transverse process. The patient's skin will be anesthetized with 2% lidocaine. A 22-gauge 10-cm needle will be inserted using an out-plane superior-to-inferior approach to place the tip into the fascial plane on the deep (anterior) aspect of erector spinae muscle. The location of the needle tip will be confirmed by visible fluid spread lifting erector spinae muscle off the bony shadow of the transverse process. A total of 30 mL of bupivacaine/lidocaine mixture will be injected.
  Arms: ESP Block
Procedure: TAP Block — TAP block will be performed at the finishing of surgery under spinal anesthesia. A linear ultrasound transducer will be placed to lateral aspect of abdomen. A 22-gauge 10-cm needle will be inserted using an out-plane superior-to-inferior approach to place the tip into the fascial plane between transversus abdominis and internal oblique muscles..A total of 30 mL of bupivacaine/lidocaine mixture will be injected.
  Arms: TAP Block
Other: Standard Pain Followup and Monitorization — Numeric Rating Scale (NRS) pain score will be recorded and followed by 0., 1.-3.-6.-12.-18.-24.hours. it is planned that the patient will continue to follow the hourly NRS score in ward. Intramuscular diclofenac will be administered in this period if NRS 4 and if it is over, intravenous 0.5 mg / kg meperidine will be administered if NRS score is 4 or more after 2 hours. Salvage analgesic needs and times will be noted in detail, and the use of rescue analgesics, as well as NRS scores at designated hours, will be kept in a statistical evaluation.
  Arms: Control; ESP Block

SUMMARY:
Multimodal analgesia is used to control postoperative pain in inguinal hernia repair. Transversus abdominis plane block is an effective regional anesthesia technique for postoperative analgesia in inguinal hernia repairs. The erector spinae plane block applied to thelow thoracic region was also reported to provide effective analgesia in these surgeries. In this study, we aimed to determine and compare the effects of transversus abdominis plane block and lumbar erector spinae plane block on postoperative pain in inguinal hernia repairs.

ELIGIBILITY:
Inclusion Criteria:

* inguinal hernia repair under spinal anesthesia, ASA 1-2-3

Exclusion Criteria:

* Patient refusal
* Contraindications to regional anesthesia
* Known allergy to local anesthetics
* Bleeding diathesis
* Use of any anti-coagulants
* Inability to provide informed consent
* Severe kidney or liver disease
* Inability to operate PCA system
* Patient with psychiatric disorders

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2018-05-10 (Actual); Study Completion 2018-05-17 (Actual)

PRIMARY OUTCOMES:
Numeric Rating Scale | 24 hours
  The numeric rating scale (NRS), the reference measurement method, will be used to determine the postoperative pain levels of the patients. Changes in NRS at rest and on movement will be recorded at intervals. NRS is a unidimensional measure of pain intensity in adults in which a respondent selects a whole number (0-10 integers) that best reflects the intensity of his/her pain. The 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable").

SECONDARY OUTCOMES:
Tramadol consumption | 24 hours
  Postoperative analgesia plan includes patient-controlled analgesia. Patient-controlled analgesia is a self-administered analgesic and a safe interval is programmed by a patient. Patients in all groups will be assessed at the end of 24 hours for tramadol consumed in patient-controlled analgesia devices.The electronic program in patient-controlled analgesia device can determine the amount of time the patient has applied the medication. The instrument's tool will be used for measurements.

CONTACTS AND LOCATIONS:
Overall Officials: serkan Tulgar, ass prof, Principal Investigator — Maltepe University
Locations (1):
- Maltepe University faculty of medicine, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Venkatraman R, Abhinaya RJ, Sakthivel A, Sivarajan G. Efficacy of ultrasound-guided transversus abdominis plane block for postoperative analgesia in patients undergoing inguinal hernia repair. Local Reg Anesth. 2016 Jan 18;9:7-12. doi: 10.2147/LRA.S93673. eCollection 2016. PMID 26848274
- [Background] Takebayashi K, Matsumura M, Kawai Y, Hoashi T, Katsura N, Fukuda S, Shimizu K, Inada T, Sato M. Efficacy of transversus abdominis plane block and rectus sheath block in laparoscopic inguinal hernia surgery. Int Surg. 2015 Apr;100(4):666-71. doi: 10.9738/INTSURG-D-14-00193.1. PMID 25875548
- [Background] Hernandez MA, Palazzi L, Lapalma J, Cravero J. Erector spinae plane block for inguinal hernia repair in preterm infants. Paediatr Anaesth. 2018 Mar;28(3):298-299. doi: 10.1111/pan.13325. Epub 2018 Jan 17. PMID 29341379